# **Document Coversheet**

Study Title: Scar Analysis in Direct Excision Brow Lift: Comparing Octyl-2- Cyanoacrylate (Dermabond) Versus Non-absorbable Sutures

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 6/18/2024 |
| NCT Number: | NCT05981443 |
| IRB Number | 88617 |
| Coversheet created: | 3/31/2025 |

0 ι co IRB Approval 6/18/2024 IRB # 88617 IRB1 CLOSED

IMPORTANT NOTE: You will not be able to change your selections for "Which IRB" and "Protocol Process Type" after having created your application. If you selected the wrong IRB or Protocol Process Type, you may need to create a new application. Please contact the Office of Research Integrity (ORI) at 859-257-9428, <a href="mailto:IRBsubmission@uky.edu">IRBsubmission@uky.edu</a>, or <a href="mailto:request a consult">request a consult</a> to resolve any questions regarding your selections.

For guidance, see:

- Which IRB?
- Which Protocol Process Type?
- "Getting Started"

| Which IRB |
|-----------------------|
| Medical |
| Protocol Process Type |
| Protocol Process Type |

The revised Common Rule expanded exemption certification category 4 for certain secondary research with identifiable information or biospecimens. The regulations no longer require the information or biospecimens to be existing. For more information see the <u>Exemption Categories Tool</u>.

#### CONTINUATION REVIEW/FINAL REVIEW

0 unresolved comment(s)

Based on your responses to the Continuation Review/Final Review questions, to be in accord with federal policy a final review report must be submitted to properly CLOSE OUT your protocol.

IF YOU WISH TO EXTEND YOUR IRB APPROVAL PERIOD, update your 'Anticipated Ending Date of Research Project' under the Project Information section and include any other supportive documentation for continuation of your study [NOTE: If you wish for your IRB approval to continue, but you do not request an extension and complete and submit your materials in a timely manner, IRB approval will expire at the end of the current approval period.].

To initiate your continuation review (CR)/annual administrative review (AAR), or properly close your study, complete this section and update/correct all other sections of your IRB application as applicable.

\*\*\*IMPORTANT\*\*\* Before leaving this page to update other sections of your application, be sure to SAVE this section first.

If you have any questions, please contact the Office of Research Integrity at 859-257-9428 or email IRBsubmission@uky.edu



## 1. Status of the Research

Check the statement(s) that best describe(s) the current status of your research: 1

- □ No subjects have enrolled to date.
- □ Recruitment and/or enrollment of new subjects or review of records/specimens continue.
- □ Study is closed to enrollment, but subjects still receive research-related interventions (e.g., treatment, blood draws).
- □ Study enrollment is permanently closed; subjects have completed all research-related interventions; and the study remains active only for long-term follow-up of subjects (see Tool Tip above for info on long-term follow-up of subjects).\*
- □ Research has progressed to the point that it involves 1) Data analysis, including analysis of identifiable private information or identifiable biospecimens; and/or 2) Accessing follow-up clinical data from procedures that subjects would undergo as part of clinical care \*
- The remaining research activities are limited only to data analysis. There is access to records or specimens either directly or through codes or links to the data.\*
- The remaining research activities are limited only to data analysis. There is no subject/record/specimen identifying codes or links to the data; the researcher or research team cannot readily ascertain the subject's identity.\*
- ☑ All study activities are complete. IRB approval can be inactivated.

# 2. If subjects have been enrolled within the last year, and the IRB approved a consent/assent form for your study:

Please attach a complete, signed copy for the last two subjects enrolled with **each** consent/assent form/HIPAA form since the last annual review.

(Example: If 3 different approved consent forms were used since the last annual review, please provide the two most recent signed copies of each version for a total of six.)

# Attachments

| Attach Type | File Name |
|----------------------------|-----------------------|
| Entire Signed Consent Form | Patient 6 consent.pdf |
| Entire Signed Consent Form | Patient 7 Consent.pdf |

## 3. Informed Consent

If the study is open to subject enrollment, please go to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- · One clean copy in PDF (without the IRB Approval stamp) of the currently approved consent/assent document(s), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is open to subject enrollment and the IRB has waived the requirement to document informed consent, please go

<sup>\*</sup>Possibility that review will move from Full to Expedited.

#### to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- One clean copy in PDF of the currently approved document used for the informed consent process (e.g., cover letter, phone script), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is closed to subject enrollment, please go to the Informed Consent section of the E-IRB Application and remove Informed Consent Documents designated to get an IRB approval stamp to avoid having them appear valid for enrollment.

## 4. Unanticipated Problems Involving Risk to Subjects or Others/Adverse Events Summary & Assessment

Did any problems/adverse events occur during the last 12 months?

In the space below, provide a written summary of both unanticipated problems\* and available information regarding adverse events since the last review (e.g., initial review or annual/continuing review). The amount of detail provided in such a summary will vary depending on the type of research being conducted; in many cases, such a summary could be a brief statement that there have been no unanticipated problems and that adverse events have occurred at the expected frequency and level of severity as documented in the research protocol, the informed consent document, and investigator's brochure (if applicable). The summary must include the Pl's assessment whether the problems/adverse events warrant changes to the protocol, consent process, or risk/benefit ratio.

Note: It is the IRB's expectation that all unanticipated problems involving risk to subjects or others or related deaths requiring prompt reporting are submitted in the appropriate time frame (See Policy [PDF]). Your response to this Annual/Continuing Review is considered assurance that all prompt reportable problems/adverse events have been submitted for IRB review.

| For multisite studies, the written summary should describe external events determined to be unanticipated problems involving risk to subjects or others. |
|---|
| 5. Subject Info To-Date |
| Our records for the previously approved IRB application indicate the <b>IRB approved estimate</b> of subjects to be enrolled (or records/specimens reviewed) is: |
| Enter the number of enrolled subjects (or records/specimens reviewed) that have not been previously reported to the IRB |
| 7 |
| Our records for the previously approved IRB application indicate the previous total # of subjects enrolled (or records/specimens reviewed) since activation of the study is: |
| The new total number of subjects enrolled (or records/specimens reviewed) since activation of the study: 7 |
| Please review the Project Info section for the IRB approved estimate of subjects to be enrolled (or records/specimens reviewed). If this new total exceeds your approved estimate of subjects to be enrolled (or records/specimens reviewed), please update the number in the field for Number of Human Subjects in the Project Info section. |

# 6. Data and Safety Monitoring Board (DSMB)/Plan (DSMP)

If your study is monitored by a DSMB or under a DSMP, attach all documentation (i.e. summary report; meeting minutes) representing Data and Safety Monitoring activities that have not been previously reported to the IRB.

Attachments

| 7. Since the most recent IRB Initial/Continuation Review Approval: | 88617<br>CLOSED |
|---|---|
| Have there been any participant complaints regarding the research? | |
| c Yes e No | |
| If yes, in the field below, provide a summary describing the complaints. | |
| Have any <b>subjects withdrawn</b> from the research voluntarily or by you as the PI for reasons related to safety, welf related to the conduct of the research? If a participant does not meet the screening criteria for a study even if they consent it is NOT considered a withdrawal. | |
| ⊂ Yes ⊚ No | |
| If yes, in the field below, provide a detailed explanation to the withdrawal(s) including if participants were lost to co | ntact. |
| Has any new and relevant literature been published since the last IRB review, especially literature relating to | risks associated with the research? |
| c Yes ⊚ No | |
| If yes, attach a copy of the literature as well as a brief summary of the literature including, if pertinent, the impact o protection of human subjects. | f the findings on the |
| Attachments | |
| Have there been any interim findings? | |
| ⊂ Yes ເ No | |
| If yes, attach a copy of Interim Findings. | |
| Attachments | |
| Have subjects experienced any benefits? | |
| ∩ Yes ເ No | |
| If yes, in the field below, provide a description of benefits subjects have experienced. | |
| Have there been any inspections/audits/quality improvement reviews of your research protocol resulting corrective action in order to protect the safety and welfare of subjects? | រូ in the need for |
| If yes, please attach documentation evidencing the outcome(s) and any corrective action(s) taken as a result | |
| Attachments | |
| Was an FDA 483 issued as a result of any inspections/audits? | |
| c Yes 6 No | |
| If yes, submit documentation using attachment button above. | |
| 8. Risk Level: | |
| Our records for the previously approved IRB application show your research is: Risk | |

# Has something during the course of your research changed the level of risk? ○ Yes ○ No

If yes, go to the Risk Level section, mark the appropriate risk level, and in the field below, describe why the risk level has changed:

## 9. Funding/Support:

Our records for the **previously approved** IRB application indicate your research is being submitted to, supported by, or conducted in cooperation with the following external or internal agency(ies) or funding program(s):

| □ Grant application pending |
|---|
| □ (HHS) Dept. of Health & Human Services |
| □ (NIH) National Institutes of Health |
| ☐ (HRSA) Health Resources and Services Administration ☐ (HRSA) Health Resources and Services Administration |
| □(DoJ) Department of Justice or Bureau of Prisons |
| □(DoE) Department of Energy |
| □ (EPA) Environmental Protection Agency |
| Federal Agencies Other Than Those Listed Here |
| □ Industry (Other than Pharmaceutical Companies) |
| □ Internal Grant Program w/ proposal |
| □ Internal Grant Program w/o proposal |
| □ National Science Foundation |
| □ Other Institutions of Higher Education |
| □ Pharmaceutical Company |
| □ Private Foundation/Association |
| □ U.S. Department of Education |
| □ State |
| Other: |

Please **update the Funding/Support section of your IRB application** if needed, including the following attachments if they contain changes not previously reported to the IRB:

- A current copy of your protocol if you are conducting industry/pharmaceutical research;
- A current Investigator Brochure (submit a copy with all changes underlined).
- · A new or revised grant application for this project.

Did your project receive extramural funding?

∩ Yes ∈ No

If yes, please review and correct if necessary, the OSPA Account # information under the **Funding/Support section** of your IRB application.

If the project is externally funded, has the sponsor offered any of the research team enrollment incentives or other personal benefit bonuses? (e.g., cash/check, travel reimbursements, gift checks, etc.)

○ Yes ○ No ⊙ N/A

Note: It is University of Kentucky policy that personal benefit bonuses are not allowed. If these conditions change during the course of the study, please notify the IRB.

# 10. Project Information

Our records for the previously approved IRB application indicate your estimated project end date is:

# 06/30/2024

If you have a new estimated project end date, please go to the Project Info section and change the date in the field for Anticipated Ending Date of Research Project.

# 11. Study Personnel

Our records for the previously approved IRB application indicate the following individuals are study personnel on this project (if applicable):

Last Name First Name

No records to display.

Please review the individuals listed above and update your records as needed in the Study Personnel section of the E-IRB application, being sure that each individual listed has completed or is up-to-date on the mandatory human research protection training [see the policy on <u>Mandatory Human Subject Protection Training FAQs</u> (required every three years)].

## 12. Progress of the Research

To meet federal requirements the IRB is relying on your RESEARCH DESCRIPTION as a protocol summary and their expectation is that it is up-to-date. If the currently approved protocol (or research description) in your E-IRB application is outdated, please make applicable changes, and describe in the field below any substantive changes and explain why they are essential. If none, insert "N/A" in the text field below. If you are closing your study, you may use the space below to summarize the final status of the research.

N/A

Note: No changes in the research procedures should have occurred without previous IRB review. Approval from the IRB must be obtained before implementing any changes.

Provide a brief summary of any modifications that affect subject safety and/or welfare approved by the IRB since the last initial or continuation review (If none, insert "N/A" in the text field below.):

N/A

Attach one copy of the most recent progress report sent to the FDA, if available. All PI-sponsored IND/IDE studies are required to submit a copy of the FDA progress report.

Attachments

# 13. Confidentiality/Security

Review your Research Description section and update the Confidentiality portion, if necessary, to describe measures for security of electronic and physical research records (e.g., informed consent document(s), HIPAA Authorization forms, sensitive or private data).

## 14. Subject Demographics

Our records for the previously approved IRB application indicate the following categories of subjects and controls are included in your research:

- ☐ Children (individuals under age 18)
- Wards of the State (Children)
- Students
- College of Medicine Students
- UK Medical Center Residents or

House Officers

- Impaired Consent Capacity Adults
- □ Pregnant Women/Neonates/Fetal

Material

- Prisoners
- Non-English Speaking
- International Citizens
- Normal Volunteers

Civilian Employees

- Patients
- Appalachian Population

Please review the Subject Demographics section of your IRB application for accuracy, and note the following:

If during the course of your research 1) any prisoners have been enrolled, OR 2) subjects have been enrolled that became involuntarily confined/detained in a penal institution that have not been previously reported to the IRB, go to Subject Demographic section in your E-IRB application and mark "prisoners" in the categories of subjects to be included in the study, if it is not already marked.

Note: If either 1 or 2 above apply, and you have received funding from the Department of Health and Human Services (HHS), a Certification Letter should have been submitted to the Office for Human Research Protections (OHRP); prisoners and individuals who have become involuntarily confined/detained in a penal institution cannot continue participation in the research until OHRP issues approval. If the Certification has not been submitted, contact the Office of Research Integrity.

Based on the total # of subjects who have enrolled, complete the subject demographic section below:

| | | Participant De | mographics | |
|---|---|---|---|---|
| | Cisgender Man 🕕 | Cisgender Woman 🗓 | TGNB/TGE 🕕 | Unknown/Not Reported |
| American _ | | | | |
| ndian/Alaskan | | | | |
| Native | | | | |
| Asian | | | | |
| Black or _ | | | | |
| African | | | | |
| American | | | | |
| Latinx | | | | |
| Native | | | | |
| Hawaiian or | | | | |
| Other Pacific | | | | |
| Islander | | | | |
| White | | | | 7 |
| American | | | | |
| Arab/Middle | | | | |
| Eastern/North L | | | | |
| African | | | | |
| Indigenous | | | | |
| People | | | | |
| Around the | | | | |
| World | | | | |
| More than | | | | |
| One Race | | | | |
| Unknown or | | | | |
| Not Reported $ot$ | | | | |

If unknown, please explain why:

Did not question gender identification

## 15. Research Sites

Our records for the previously approved IRB application indicate that you are conducting research at the following sites:

UK Sites

■ UK Classroom(s)/Lab(s)

**■ UK Healthcare Good Samaritan Hospital** 

| ⊏ UK Hospital |
|---|
| Schools/Education Institutions Schools/Education Institutions |
| □ Fayette Co. School Systems * |
| ■ Other State/Regional School Systems |
| □ Institutions of Higher Education (other than UK) |
| Other Medical Facilities |
| □ Bluegrass Regional Mental Health Retardation Board □ Cardinal Hill Hospital |
| ☐ Eastern State Hospital |
| □ Nursing Homes |
| ☐ Shriner's Children's Hospital ☐ Shriner's Children's Hospital ☐ Shriner's Children's Hospital ☐ Shriner's Children's Hospital ☐ Shriner's Children's Hospital |
| ☐ Other Hospitals and Med. Centers |
| Correctional Facilities |

If the above listed sites are not accurate, go to the Research Sites section of the E-IRB application to update the facilities at which

If you are adding a new off-site facility, you may also need to update your E-IRB application Research Description, Research Sites, Informed Consent, and other affected sections as well as any documents which will list the off-site facility. Documents needing updating may include, but not limited to:

- · Consent forms (attachment under Informed Consent section)
- Brochures (attachment under Additional Info section)

research procedures have been or will be conducted.

- Advertisements (attachment under Research Description section);
- Letter of support (attachment under Research Sites section)).

Please revise applicable sections and attachments as necessary.

# 16. Disclosure of Significant Financial Interest

☐ Home Health Agencies
☐ International Sites

Other:

Disclosure of Significant Financial Interest:

Our records for the previously approved IRB application indicate that you, your investigators, and/or key personnel (KP) have a significant financial interest (SFI) related to your/their responsibilities at the University of Kentucky (that requires disclosure per the UK administrative regulation 7:2):

If you need to update your records, please go to the PI Contact Information section and/or Details for individuals listed in the Study Personnel section to change your response to the applicable question(s).

## 17. Supplementals

To ensure the IRB has the most accurate information for your protocol you are expected to re-visit the E-IRB application sections and make corrections or updates as needed. At a minimum you are being asked to review the following sections for accuracy:

STUDY DRUG INFORMATION—Please review for accuracy. STUDY DEVICE INFORMATION—Please review for accuracy. RESEARCH ATTRIBUTES—Please review for accuracy. OTHER REVIEW COMMITTEES -- Please review for accuracy.

# **PROJECT INFORMATION**

0 unresolved comment(s)

Title of Project: (Use the exact title listed in the grant/contract application, if applicable). If your research investigates any aspect of COVID-19, please include "COVID19" at the beginning of your Project Title and Short Title Scar analysis in direct excision brow lift: comparing octyl-2-cyanoacrylate (Dermabond) versus non-absorbable sutures

Short Title Description

Please use a few key words to easily identify your study - this text will be displayed in the Dashboard listing for your study.

Brow Lift Scar Analysis

Anticipated Ending Date of Research Project: 6/30/2024

Maximum number of human subjects (or records/specimens to be reviewed) 40

After approval, will the study be open to enrollment of new subjects or new data/specimen collection? 6 Yes No

Are you requesting that the UK IRB serve as the lead IRB for a multi-site study, OR that the UK IRB defer review to another IRB? [Click here for "IRB Reliance" help]

Yes 6 No

If "Yes," before completing your IRB application, fill out the Reliance Request Form and submit it to irbreliance@uky.edu.

## PI CONTACT INFORMATION

0 unresolved comment(s)

## Principal Investigator (PI) role for E-IRB access

The PI is the individual holding primary responsibility on the research project with the following permissions on the E-IRB application:

- 1. Read;
- 2. write/edit;
- 3. receive communications; and
- 4. submit to the IRB (IR, CR, MR, Other Review\*).

If research is being submitted to or supported by an extramural funding agency such as NIH, a private foundation or a pharmaceutical/manufacturing company, the PI listed on the grant application or the drug protocol must be listed as PI here.

Please fill in any blank fields with the appropriate contact information (gray shaded fields are not editable). Required fields left blank will be highlighted in pink after you click "Save".

To change home and work addresses, go to <a href="myUK">myUK</a> and update using the Employee Self Service (ESS) portal. If name has changed, the individual with the name change will need to submit a <a href="mailto:">Name Change Form</a>' to the Human Resources Benefits Office for entering into SAP. The new name will need to be associated with the individual's Link Blue ID in SAP before the change is reflected in E-IRB. Contact the <a href="https://example.com/HR Benefits">HR Benefits Office</a> for additional information.

The Principal Investigator's (PI) contact information is filled in automatically based on who logged in to create the application.

#### If you are not the Principal Investigator, do NOT add yourself as study personnel.

To change the PI contact information on an application in Researcher edit status:

- click "Change Principal Investigator";
- search for the PI's name using the search feature;
- click "Select" by the name of the Principal Investigator, then "Save Contact Information".

You will automatically be added as study personnel with editing permissions to continue editing the application.



## **Change Principal Investigator:**

| First Name | | Room# & | |
|---|---|---|---|
| First Name: | Peter | Bldg: E320 | KY CLINIC |
| Last Name: | Timoney | <u>Speed</u><br><u>Sort#</u> : 1 40536 | 60284 |
| Middle Name | John | | |
| Department: | Ophthalmology & Visual Scie | Dept Code: 7H85 | 4 |
| Pl's | | Rank: 🕕 | |
| Employee/Student<br>ID#: | 00033583 | | Associate Professor |
| PI's Telephone #: | N/A | Degree: | MD |
| Pl's e-mail<br>address: | pjtimo2@uky.edu | PI's FAX<br>Number: | |
| PI is R.N. 🛈 | ⊂ Yes ເ No | HSP Trained: | Yes |
| | | HSP Trained<br>Date: | 8/25/2021 |
| | | RCR Trained: | Yes |
| | a <u>significant financial interest</u> related t<br><u>Kadministrative regulation 7:2</u> )? | to your responsibilities at the U | niversity of Kentucky (that requires |

RISK LEVEL 0 unresolved comment(s)

Indicate which of the categories listed below accurately describes this protocol

- (Risk Level 1) Not greater than minimal risk
- ¬ (Risk Level 2) Greater than minimal risk, but presenting the prospect of direct benefit to individual subjects.
- െ (Risk Level 3) Greater than minimal risk, no prospect of direct benefit to individual subjects, but likely to yield generalizable knowledge about the subject's disorder or condition.
- \*"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves from those ordinarily encountered in daily life or during the performance of routine physical or psychological examination or tests.

Refer to <u>UK's guidance document</u> on assessing the research risk for additional information.



0 unresolved comment(s)

#### SUBJECT DEMOGRAPHICS

Age level of human subjects: (i.e., 6 mths.; 2yrs., etc..) 18 to 100

#### Study Population:

Describe the characteristics of the subject population, including age range, gender, ethnic background and health status. Identify the criteria for inclusion and exclusion.

Provide the following information:

- · A description of the subject selection criteria and rationale for selection in terms of the scientific objectives and proposed study design;
- A compelling rationale for proposed exclusion of any sex/gender or racial/ethnic group;
- Justification for the inclusion of vulnerable groups such as children, prisoners, adults with impaired consent capacity, or others who may be vulnerable to coercion or undue influence.

Please consider these resources:

**NIH Diversity Policy** 

FDA Diversity Guidance 10

Subjects will consist of UK Oculoplastics patients found to have brow ptosis in need of surgical repair. There will be no vulnerable groups included in our study population, nor will any specific gender, racial, or ethnic groups be excluded.

#### Inclusion criteria:

- -Patients undergoing bilateral direct excision brow lift for brow ptosis at the University of Kentucky Medical Center.
- -Patients > 18 years of age
- -Patients must be able to follow up at the specified intervals.
- -Patients who are able to give their own informed consent.
- -Health Status: Variable health status reflective of general population of Kentucky. Patients will be healthy enough to be seen in an office setting.
- -No patient will be excluded on the basis of gender, ethnicity, or religious background.
- -All patients will need to be proficient in the English language to understand the scale used for scar assessment

#### Exclusion Criteria:

- -Patients <18 years of age or >100
- -Allergy to octyl-2-cyanoacrylate
- -Adults with impaired consent capacity
- -Incarcerated individuals

#### Attachments

Indicate the targeted/planned enrollment of the following members of minority groups and their subpopulations. Possible demographic sources: Census Regional Analyst Edition, Kentucky Race/Ethnic Table, Kentucky Population Data.

(Please note: The IRB will expect this information to be reported at Continuation Review time for Pre-2019 FDA-regulated Expedited review and Full review applications):

| | | Participant Demo | graphics | |
|---|---|---|---|---|
| | Cisgender Man 🛈 | Cisgender Woman 🗓 | TGNB/TGE 🕡 | Unknown/Not Reported |
| American | | | | |
| Indian/Alaskan | | | | |
| Native: | | | | |
| Asian: | | | | |
| Black/African | | | | |
| American: | | | | |
| Latinx: | | | | |
| Native | | | | |
| awaiian/Pacific | | | | |
| Islander: | | | | |
| White: | | | | |
| American | | | | |
| Arab/Middle | | | | |
| Eastern/North | | | | |
| African: | | | | |
| Indigenous | | | | |
| People Around the World: | | | | |
| More than One | | | | |
| Race: | | | | |
| Jnknown or Not | | | | |
| Reported: | | | | |



This will vary based on the identification of the patient population that present to the UK Oculoplastics clinics. We will not recruit or discriminate by ethnicity.

Indicate the categories of subjects and controls to be included in the study. You may be required to complete additional forms depending on the subject categories which apply to your research. If the study does not involve direct intervention or direct interaction with subjects, (e.g., record-review research, outcomes registries), do not check populations which the research does not specifically target. For example: a large record review of a diverse population may incidentally include a prisoner or an international citizen, but you should not check those categories if the focus of the study has nothing to do with that status.

Check All That Apply (at least one item must be selected)

## ADDITIONAL INFORMATION:

□ Children (individuals under age 18)

- □ Wards of the State (Children)
- □ Emancipated Minors
- ☐ Students
- □ College of Medicine Students
- □ UK Medical Center Residents or House Officers
- □ Impaired Consent Capacity Adults
- □ Pregnant Women/Neonates/Fetal Material
- □Prisoners
- ☐ Non-English Speaking (translated long or short form)
- □ International Citizens
- □ Normal Volunteers
- ☐ Military Personnel and/or DoD Civilian Employees
- ☑ Patients
- □ Appalachian Population

Please visit the <u>IRB Survival Handbook</u> for more information on:

- Children/Emancipated Minors
- Students as Subjects
- Prisoners
- Impaired Consent Capacity Adults
- Economically or Educationally Disadvantaged Persons

## Other Resources:

- UKMC Residents or House Officers [see requirement of GME]
- Non-English Speaking [see also the E-IRB Research Description section on this same topic]
- International Citizens [DoD SOP may apply]
- Military Personnel and/or DoD Civilian Employees

# Assessment of the potential recruitment of subjects with impaired consent capacity (or likelihood):

Check this box if your study does NOT involve direct intervention or direct interaction with subjects (e.g., record-review research, secondary data analysis). If there is no direct intervention/interaction you will not need to answer the impaired consent capacity questions.

Does this study focus on adult subjects with any conditions that present a high *likelihood* of impaired consent capacity or *fluctuations* in consent capacity? (see examples below)

If Yes and you are not filing for exemption certification, go to "Form T", complete the form, and attach it using the button below.

## Examples of such conditions include:

- Traumatic brain injury or acquired brain injury
- Severe depressive disorders or Bipolar disorders
- Schizophrenia or other mental disorders that
- involve serious cognitive disturbances
- Stroke
- Developmental disabilities
- Degenerative dementias
- CNS cancers and other cancers with possible CNS involvement
- Late stage Parkinson's Disease

- Late stage persistent substance dependence
- Ischemic heart disease
- HIV/AIDS
- COPD
- · Renal insufficiency
- Diabetes
- Autoimmune or inflammatory disorders
- Chronic non-malignant pain disorders
- Drug effects
- Other acute medical crises



## INFORMED CONSENT/ASSENT PROCESS/WAIVER

0 unresolved comment(s)

For creating your informed consent attachment(s), please download the most up-to-date version listed in "All Templates" under the APPLICATION LINKS menu on the left, and edit to match your research project.

#### Additional Resources:

- Informed Consent/Assent Website
- Waiver of Consent vs. Waiver of Signatures
- Sample Repository/Registry/Bank Consent Template

## Consent/Assent Tips:

- If you have multiple consent documents, be sure to upload each individually (not all in a combined file).
- If another site is serving as the IRB for the project, attach the form as a "Reliance Consent Form" so the document will not receive a UK IRB approval stamp; the reviewing IRB will need to stamp the consent forms.
- Changes to consent documents (e.g., informed consent form, assent form, cover letter, etc...) should be reflected in a 'tracked changes' version and uploaded separately with the Document Type "Highlighted Changes".
- It is very important that only the documents you wish to have approved by the IRB are attached; DELETE OUTDATED FILES -previously approved versions will still be available in Protocol History.
- Attachments that are assigned a Document Type to which an IRB approval stamp applies will be considered the version(s) to be
  used for enrolling subjects once IRB approval has been issued.
   Document Types that do NOT get an IRB approval stamp are:
  - · "Highlighted Changes",
  - · "Phone Script", and
  - · "Reliance Consent Form",
  - "Sponsor's Sample Consent Form".

#### How to Get the Section Check Mark

- 1. You must:
  - a) provide a response in the text box below describing how investigators will obtain consent/assent, and
  - b) check the box for at least one of the consent items and/or check mark one of the waivers
- 2. If applicable attach each corresponding document(s) as a read-only PDF.
- 3. If you no longer need a consent document approved (e.g., closed to enrollment), or, the consent document submitted does not need a stamp for enrolling subjects (e.g., umbrella study, or sub-study), only select "Stamped Consent Doc(s) Not Needed".
- 4. After making your selection(s) be sure to scroll to the bottom of this section and SAVE your work!



#### Check All That Apply

- ☐ Assent Form
- ☐ Cover Letter (for survey/questionnaire research)
- □ Phone Script
- □ Informed Consent/HIPAA Combined Form
- □ Debriefing and/or Permission to Use Data Form
- □ Reliance Consent Form
- □ Sponsor's sample consent form for Dept. of Health and Human Services (DHHS)-approved protocol
- ☐ Stamped Consent Doc(s) Not Needed



# Informed Consent Process:

Using active voice, describe how investigators will obtain consent/assent. Include:

- the circumstances under which consent will be sought and obtained
- · the timing of the consent process (including any waiting period between providing information and obtaining consent)

- · who will seek consent
- how you will minimize the possibility of coercion or undue influence
- the method used for documenting consent
- if applicable, who is authorized to provide permission or consent on behalf of the subject
- if applicable, specific instruments or techniques to assess and confirm potential subjects' understanding of the information

Note: all individuals authorized to obtain informed consent should be designated as such in the E-IRB "Study Personnel" section of this application.

Special considerations may include:

- · Obtaining consent/assent for special populations such as children, prisoners, or people with impaired decisional capacity
- Research Involving Emancipated Individuals
   If you plan to enroll some or all prospective subjects as emancipated, consult with UK legal counsel prior to submitting this application to the IRB. Include research legal counsel's recommendations in the "Additional Information" section as a separate document
- Research Involving Non-English Speaking Subjects
   For information on inclusion of non-English speaking subjects, or subjects from a foreign culture, see IRB Application Instructions for Recruiting Non-English Speaking Participants or Participants from a Foreign Culture.
- Research Repositories
   If the purpose of this submission is to establish a research repository describe the informed consent process. For guidance regarding consent issues, process approaches, and sample language see the <a href="Sample Repository/Registry/Bank Consent Template">Sample Repository/Registry/Bank Consent Template</a>.

The patients will be consented for the study once a determination has been made that they are surgical candidates. This will occur in the clinic after describing the study. Consent will be obtained preferably by research coordinators in the Ophthalmology department that have no role in patient care, but if necessary due to lack of staffing or availability, by residents, fellows, or attendings in the UK Oculoplastics clinic. Patients will be assured that their choice to participate or not in the study will have no bearing on their surgical experience and they are free to decline to participate and receive the current standard of care procedure involving suturing. The consent forms will be stored under lock and key in the PI's office, and if electronic copies are made, they will be stored in encrypted servers using a file storage provider contracted through the University of Kentucky.

□ Request for Waiver of Informed Consent Process

If you are requesting IRB approval to waive the requirement for the informed consent process, or to alter some or all of the elements of informed consent, complete, Section 1 and Section 2 below.

Note: The IRB does not approve waiver or alteration of the consent process for greater than minimal risk research, except for planned emergency/acute care research as provided under FDA regulations. Contact ORI for regulations that apply to single emergency use waiver or acute care research waiver (859-257-9428).

## **SECTION 1.**

Check the appropriate item:

■I am requesting a waiver of the requirement for the informed consent process.

■I am requesting an alteration of the informed consent process.

If you checked the box for this item, describe which elements of consent will be altered and/or omitted, and justify the alteration.

# SECTION 2.

Explain how each condition applies to your research.

- a) The research involves no more than minimal risk to the subject.
- b) The rights and welfare of subjects will not be adversely affected.
- c) The research could not practicably be carried out without the requested waiver or alteration.
- d) Whenever possible, the subjects or legally authorized representatives will be provided with additional pertinent information after they have participated in the study.
- e) If the research involves using or accessing identifiable private information or identifiable biospecimens, the research could not practicably be carried out without using such information or biospecimens in an identifiable format.
  - Private information/specimens are "identifiable" if the investigator may ascertain the identity of the subject or if identifiers
    are associated with the information (e.g., medical records). This could be any of the <u>18 HIPAA identifiers</u> including <u>dates</u>
    of service.
  - If not using identifiable private information or identifiable biospecimens, insert N/A below.

If you are requesting IRB approval to waive the requirement for signatures on informed consent forms, **your research** activities must fit into one of three regulatory options:

- 1. The only record linking the participant and the research would be the consent document, and the principal risk would be potential harm resulting from a breach of confidentiality (e.g., a study that involves participants who use illegal drugs).
- 2. The research presents no more than minimal risk to the participant and involves no procedures for which written consent is normally required outside of the research context (e.g., a cover letter on a survey, or a phone script).
- 3. The participant (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm, the research presents no more than minimal risk to the subject, and there is an appropriate alternative mechanism for documenting that informed consent was obtained.

Select the option below that best fits your study.

If the IRB approves a waiver of signatures, participants must still be provided oral or written information about the study. To ensure you include required elements in your consent document, use the **Cover Letter Template** as a guide. There is an English and a Spanish version.



# © Option 1

## Describe how your study meets these criteria:

- a) The only record linking the participant and the research would be the consent document:
- b) The principal risk would be potential harm resulting from a breach of confidentiality (i.e., a study that involves subjects who use illegal drugs).

Under this option, each participant (or legally authorized representative) must be asked whether (s)he wants to sign a consent document; if the participant agrees to sign a consent document, only an IRB approved version should be used.

#### Option 2

## Describe how your study meets these criteria:

- a) The research presents no more than minimal risk to the participant:
- b) Involves no procedures for which written consent is normally required outside of the research context (i.e. a cover letter on a survey, or a phone script):

## Option 3

## Describe how your study meets these criteria:

- a) The subject (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm.
- b) The research presents no more than minimal risk to the subject.
- c) There is an appropriate alternative mechanism for documenting that informed consent was obtained.

STUDY PERSONNEL 0 unresolved comment(s)

Do you have study personnel who will be assisting with the research?

After selecting 'Yes' or 'No' you must click the 'Save Study Personnel Information' button.

Yes c No

## Manage Study Personnel

Identify other study personnel assisting in research project:

- The individual listed as PI in the 'PI Contact Information' section should NOT be added to this section.
- If the research is required for a University of Kentucky academic program, the faculty advisor is also considered study personnel and should be listed below.
   \*\*\*Residents and students who are PI's are encouraged to designate the faculty advisor or at least one other individual as a contact with an editor role (DP).
- Role: DP = Editor (individual can view, navigate, and edit the application for any review phase (IR, CR/FR, MR) or 'Other Review", and submit Other Reviews on behalf of the PI.)
- Role: SP = Reader (individual can view and navigate through the currently approved application only.)

To add an individual via the below feature:

- · Search for personnel;
- · Click "select" by the listing for the person you want to add;
- For each person, specify responsibility in the project, whether authorized to obtain informed consent, AND denote who should receive E-IRB notifications (contact status).

NOTE: Study personnel must complete human subject protection (HSP) and Responsible Conduct of Research (RCR) training before implementing any research procedures. For information about training requirements for study personnel, visit UK's <u>HSP FAQ page</u>, the <u>RCR Getting Started page</u>, or contact ORI at 859-257-9428. If you have documentation of current HSP training other than that acquired through UK CITI, you may submit it to ORI (<u>HSPTrainingSupport@uky.edu</u>) for credit.

Study personnel assisting in research project: 0

| Last<br>Name | First<br>Name | Responsibility<br>In Project | Role | A<br>C | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | Last<br>Updated | SFI | Active |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Blanchard | Cody | Co-<br>Investigator | DP | N | Υ | MD | Р | Υ | 10/05/2022 | Υ | N | 06/07/2023 | N | Υ |
| Dampier | Connie | Study<br>Coordinator | DP | Υ | Υ | | Р | Υ | 06/17/2024 | Υ | N | 06/07/2023 | N | Υ |
| Gupta | Lalita | Co-<br>Investigator | DP | Υ | Υ | MD | Р | Υ | 10/19/2022 | Υ | N | 06/07/2023 | N | Υ |
| James | Yvonne | Study<br>Coordinator | DP | Υ | N | | Р | Υ | 04/14/2023 | Υ | N | 07/18/2023 | N | Υ |
| Kuhl | Sara | Study<br>Coordinator | DP | Υ | Υ | | Р | Υ | 08/10/2023 | Υ | N | 06/07/2023 | N | Υ |

## RESEARCH DESCRIPTION

0 unresolved comment(s)

You may attach a sponsor's protocol pages in the "Additional Information" section and refer to them where necessary in the Research Description. However, each prompt that applies to your study should contain at least a summary paragraph.

## Pro Tips:

- Save your work often to avoid losing data.
- Use one of the attachment buttons in this section or under the Additional Information section to include supplemental
  information with your application. During the document upload process, you will be able to provide a brief description
  of the attachment.

#### Background

Include a brief review of existing literature in the area of your research. You should identify gaps in knowledge that should be addressed and explain how your research will address those gaps or contribute to existing knowledge in this area. For interventional research, search PubMed and ClinicalTrials.gov for duplicative ongoing and completed trials with same condition and intervention(s).

Eyebrow ptosis commonly occurs with age and can result in significant patient distress with decreased visual fields, compromised activities of daily living, and aesthetic concerns. Operations to correct the ptotic brow date back to the early 1900's. Passot described excision of the skin and soft tissue directly above the lateral brow in 1930 and it has remained as a popular technique. Alternative procedures include coronal incision with lift, mid-forehead lift, and endoscopic brow lifts. The direct excision brow lift allows clear visualization of adjustments made in brow position and the impact on surrounding facial landmarks. It is also relatively quick and straightforward but it is often criticized for an unsightly facial scar. However, with proper skin closure techniques, studies have shown adequate patient satisfaction with their outcomes.

Given the prominent location of these scars and the associated social stigma, we feel it is important to focus on the skin closure methods. Skin closure is a critical portion of the operation and may be performed with sutures, skin glue, or staples. A trend has evolved utilizing skin glue (octyl-2-cyanoacrylate, Dermabond®) as it is thought to be faster, leading to shorter operating room times, potentially less cost, less risk for needle stick injuries, provides barrier to contamination, and does not require the sometimes painful suture removal. Sutures are thought to take more operating room time and require removal in outpatient clinic. There is also more variability with surgeon technique. Greene et al (1999) performed a study with the much thinner skin of the upper eyelids in blepharoplasties and found equivalent results in scar appearance, complications, and patient satisfaction. However, a Cochrane review to comparing tissue adhesives to skin glue found the latter actually took more time and was associated with more wound dehiscence. No studies looked at the use of these adhesives in the direct excision brow lift.

In terms of monetary expenditures, one tube of octyl-2-cyanoacrylate costs approximately \$24. Macario et al site that one minute of operating room time costs approximately \$29, varying in case complexity. We would like to assess the total costs between the two techniques when time in the OR is taken into account.

We hypothesize that the scars will be equivalent in assessment and ultimately be less costly with less patient distress. We also suspect that the skin glue may create an occlusive barrier to infectious contamination of the wounds and potentially a lower complication rate.

## **Objectives**

List your research objectives. Please include a summary of intended research objectives in the box below.

- 1. To determine if octyl-2-cyanoacrylate provides equivalent wound healing compared to conventional non-absorbable skin suture techniques
- 2. To determine if octyl-2-cyanoacrylate provides equivalent scar appearance compared to conventional non-absorbable suture techniques
- 3. To determine the cost effectiveness of the use of octyl-2-cyanoacrylate for skin closure compared to conventional non-absorbable suture techniques
- 4. To determine if octyl-2-cyanoacrylate results in equivalent complication rates compared to conventional non-absorbable suture techniques

#### Study Design

Describe and explain the study design (e.g., observational, secondary analysis, single/double blind, parallel, crossover, deception, etc.).

- · Clinical Research: Indicate whether subjects will be randomized and whether subjects will receive any placebo.
- Community-Based Participatory Research: If you are conducting community-based participatory research (CBPR), describe
  strategies for involvement of community members in the design and implementation of the study, and dissemination of results from
  the study.
- Qualitative research: Indicate ranges where flexibility is needed, if a fixed interview transcript is not available, describe interview topics including the most sensitive potential questions.

Research Repositories: If the purpose of this submission is to establish a Research Repository (bank, registryou plan to collect is already available from a commercial supplier, clinical lab, or established IRB approved research repository, provide scientific justification for establishing an additional repository collecting duplicate material. Describe the repository design and operating procedures. For relevant information to include, see the <u>UK Research Biospecimen Bank Guidance</u> or the <u>UK Research Registry Guidance</u>.

The proposed study is a two staged prospective study comparing skin closure with octyl-2-cyanoacrylate (Dermabond) with conventional non-absorbable sutures in the direct excision brow lift.

In stage 1, subjects will be consented to receive one of two surgical closing techniques on a bilateral brow ptosis repair: 1) deep dermal sutures and superficial interrupted sutures (the standard of care at the University of Kentucky); or 2) deep dermal sutures and octyl-2-cyanoacrylate skin glue application for superficial closing. Subjects will undergo a single closing technique on both sides. Four subjects will complete surgery in each arm (n=8 subjects total: n=4 for arm 1, and n=4 for arm 2). After the follow-up period, the scar appearance between groups will be compared. If there the octyl-2-cyanoacrylate (dermabond) group have worse appearing scars, then we will not continue to study. If the difference in appearance is negligible, then we will return to the IRB for approval to advance to stage two.

#### Stage two is outlined below:

Each patient will serve as their own control, with one brow undergoing skin closure with interrupted 6-0 prolene suture and the other with octyl-2-cyanoacrylate skin glue. Deep dermal sutures will placed in both wounds at 1 cm intervals. The patients will be randomized as to which side receives what type of closure (i.e. the right side receiving skin glue and the left receiving skin sutures or vice versa). This will prevent acquired bias during the scar analysis. The operation is done under monitored anesthesia care. We will record the time it takes to close both wounds. We will determine the precise costs of the skin glue and suture and the incurred costs per minute of operating room time. We will monitor the patients after discharge for any complications (infection, wound dehiscence, skin reaction, etc), which will be recorded. Patients will follow up at 10 days, and 3 months. Photos will be taken at the follow up visits with patient's consent. The scars will be aesthetically analyzed by plastic surgeons in terms of which scar is more aesthetically pleasing. In addition, the patient and observer (physician) will analyze the scar using the well established Patient and Observer Scar Assessment Scale. The physicians completing the forms are the research personnel.

## Attachments

#### Subject Recruitment Methods & Advertising

Describe how the study team will identify and recruit subjects. Please consider the following items and provide additional information as needed so that the IRB can follow each step of the recruitment process.

- How will the study team identify potential participants?
- · Who will first contact the potential subjects, and how?
- Will you use advertisements? If so, how will you distribute those?
- How and where will the research team meet with potential participants?
- If applicable, describe proposed outreach programs for recruiting women, minorities, or disparate populations.
- How you will minimize undue influence in recruitment?
- · Attach copies of all recruiting and advertising materials (emails, verbal scripts, flyers, posts, messages, etc.).

For additional information on recruiting and advertising:

- IRB Application Instructions Advertisements
- PI Guide to Identification and Recruitment of Human Subjects for Research

Patient participants will be recruited from University of Kentucky Oculoplastics clinic setting. They will undergo a thorough history and physical examination and carry a diagnosis of bilateral brow ptosis. If they meet the inclusion criteria and are found to be appropriate for the study, enrollment will be discussed. The investigators will obtain a formal informed consent.

# Attachments

#### Research Procedures

Describe how the research will be conducted.

- What experience will study participants have?
- What will study participants be expected to do?
- How long will the study last?
- Outline the schedule and timing of study procedures.
- Provide visit-by-visit listing of all procedures that will take place.
- Identify all procedures that will be carried out with each group of participants.
- Describe deception and debrief procedures if deception is involved.

Differentiate between procedures that involve standard/routine clinical care and those that will be performed specifically for this research project. List medications that are explicitly forbidden or permitted during study participation.

Informed consent will be obtained prior to enrollment in the study. The patient will undergo thorough history and physical examination in the clinic setting. We will then schedule for surgery if all criteria are met. The anesthesia staff will administer the standard and appropriate anesthetic. Local anesthesia will be administered. For step one of this research project the surgical procedure will be identical for all patients except the final superficial skin closure. We will design the amount of upper lateral superior brow tissue requiring excision to correct the patient's ptosis. Calipers will be used to ensure precise measurements. We will use a 15 blade to incise through the skin to the level of the frontalis muscle and fascia on both sides. Hemostasis will be achieved with Bovie electrocautery over the wounds. Both brows will be closed with 5-0 Vicryl in the subcutaneous and deep dermal layers spaced at 1 cm apart. The skin layer will be closed using interrupted 6-0 prolene sutures or with octyl-2-cyanoacrylate bilaterally. Patients will be randomized into either group. Photos will be taken both before the procedure and afterwards for research purposes. Then an independent group will evaluate photos and scar surveys for acceptability of results. The group will prepare a summary report. The photos and the summary report will be submitted to the IRB. If the the 6-0 prolene closure technique and octyl-2-cyanoacrylate closure technique are deemed to be equivocal, a request to move to Phase 2 will be made.

In phase 2 of the research project, a group of patients will all undergo the same procedure but each patient will be their own control. One side will be closed with interrupted 6-0 proline sutures and the other side closed with octyl-2-cyanoacrylate, it will be randomized what side will get which superficial skin closure.

Attachments

#### **Data Collection & Research Materials**

In this section, please provide the following:

- Describe all sources or methods for obtaining research materials about or from living individuals (such as specimens, records, surveys, interviews, participant observation, etc.), and explain why this information is needed to conduct the study.
- For each source or method described, please list or attach all data to be collected (such as genetic information, interview scripts, survey tools, data collection forms for existing data, etc.).
- If you will conduct a record or chart review, list the beginning and end dates of the records you will view.

See attachments for the POSAS survey that will be used to grade scar appearance.

# Attachments

| Attach Type | File Name |
|----------------|---------------------------------------------|
| DataCollection | 77074_DataCollection_267377.pdf |
| DataCollection | dss_2017_12_22_patel_ds-00686-2016_sdc1.pdf |

# Resources

Describe the availability of the resources and adequacy of the facilities that you will use to perform the research. Such resources may include:

- Staffing and personnel, in terms of availability, number, expertise, and experience;
- Computer or other technological resources, mobile or otherwise, required or created during the conduct of the research;
- Psychological, social, or medical services, including equipment needed to protect subjects, medical monitoring, ancillary care, or counseling or social support services that may be required because of research participation;
- Resources for communication with subjects, such as language translation/interpretation services.

Patient histories, physical examinations, and discussions regarding candidacy for the study will occur in the University of Kentucky Ophthalmology Clinics. The operations will be performed at the University of Kentucky Center for Advanced Surgery. The equipment used to perform the procedure will be in accordance with the usual standard of care for a direct excision brow lift. Dr. Timoney and the enrolled patient will fill out the described questionnaires. We do not anticipate the need for psychological or social services. We do not anticipate the need for special medical monitoring, ancillary care, equipment needed to protect subject other the usual standards in perioperative and intraoperative care.

#### Potential Risks & Benefits

#### Risks

- Describe any potential risks including physical, psychological, social, legal, ability to re-identify subjects, or other risks. Assess
  the seriousness and likelihood of each risk.
- Which risks may affect a subject's willingness to participate in the study?
- · Describe likely adverse effects of drugs, biologics, devices or procedures participants may encounter while in the study.
- Qualitative research describe ethical issues that could arise while conducting research in the field and strategies you may use to handle those situations.
- Describe any steps to mitigate these risks.

## Benefits

- Describe potential direct benefits to study participants including diagnostic or therapeutic, physical, psychological or emotional, learning benefits. This cannot include incentives or payments.
- · State if there are no direct benefits.
- Describe potential benefits to society and/or general knowledge to be gained.

Describe why potential benefits are reasonable in relation to potential risks. If applicable, justify why risks to vulnerable subjects are reasonable to potential benefits.

Potential skin reactions to octyl-2-cyanoacrylate, Dermabond®, have been described but are rare. If patients have a known allergy, they will be excluded from the study. To avoid potential complications of dehiscence, we will be placing deep dermal sutures in addition to both superficial skin closures. Another risk is the possible, but unlikely, breach of confidentiality.

Direct excision brow lifts improve patient visual fields allowing them the better engage in activities of daily living. The prominent location of the scar is concerning for many patients and carries a social stigma. Therefore, determining the most aesthetic closure technique may improve patients' quality of life. In addition, we will determine the cost benefit of each technique. Neither method imposes any significant risk the patient. They are widely used techniques but have not been compared for direct brow lifts.

## Available Alternative Opportunities/Treatments

Describe alternative treatments or opportunities that might be available to those who choose not to participate in the study, and which offer the subject equal or greater advantages. If applicable, this should include a discussion of the current standard of care treatment(s).

Both skin closure methods discussed above are in compliance with the current standard of care. If patients decide not to enroll in the study, they will undergo a two to three layer suture closure with the same closure on both sides. In addition, photos for research purposes will not be taken and questionnaires will not be distributed.

Back to Top

# Records, Privacy, and Confidentiality

Specify where the data and/or specimens will be stored and how the researcher will ensure the privacy and confidentiality of both. Specify who will have access to the data/specimens and why they need access.

Describe how data will be managed after the study is complete:

- If data/specimens will be maintained, specify whether identifiers will be removed from the maintained information/material.
- If identifiers will not be removed, provide justification for retaining them and describe how you will protect confidentiality.
- If the data/specimens will be destroyed, verify that this will not violate <u>retention policies</u> and will adhere to applicable facility requirements.

If this study will use de-identified data from another source, describe what measures will be taken to ensure that subject identifiers are not given to the investigator.

If applicable, describe procedures for sharing data/specimens with collaborators not affiliated with UK.

For additional considerations:

Return of Research Results or Incidental Research Findings

**HIPAA** policies

FERPA policies

Procedures for Transfer agreements

Information regarding multi-site studies

NIH Genomic Data Sharing (GDS) Policy

Digital Data

The obtained information will be de-identified and stored by a unique subject number (001, 002, etc.). It will be stored on an Excel sheet and in files on a password protected computer in the locked investigator's office at the University of Kentucky. Only the

investigators listed on the IRB will have access to this information. Six years after the studies conclusion, the data according to University of Kentucky policy.

<u>UK IRB policies</u> state that IRB-related research records must be retained for a minimum of 6 years after study closure. Do you confirm that you will retain all IRB-related records for a minimum of 6 years after study closure?

• Yes • No

## **Payment**

Describe the incentives (monetary or other) being offered to subjects for their participation. If monetary compensation is offered, indicate the amount and describe the terms and schedule of payment. Please review <a href="mailto:this guidance">this guidance</a> for more information on payments to subjects, including restrictions and expectations.

There will be no payment or compensation.

#### Costs to Subjects

Include a list of services and/or tests that will not be paid for by the sponsor and/or the study (e.g., MRI, HIV). Keep in mind that a subject will not know what is "standard" – and thus not covered by the sponsor/study – unless you tell them.

Both skin closure techniques involved in the study are consistent with the current standard of care. We are comparing two techniques commonly used by practicing surgeons. Because the surgeon could select either closure technique in the operation in a non- research setting, these are not considered additional costs.

#### **Data and Safety Monitoring**

The IRB requires review and approval of data and safety monitoring plans for greater than minimal risk research or NIH-funded/FDA-regulated clinical investigations.

- If you are conducting greater than minimal risk research, or your clinical investigation is NIH-funded, describe your Data and Safety Monitoring Plan (DSMP). <u>Click here for additional guidance on developing a Data and Safety Monitoring Plan</u>.
- If this is a non-sponsored investigator-initiated protocol considered greater than minimal risk research, and if you are planning on using a Data and Safety Monitoring Board (DSMB) as part of your DSMP, <u>click here for additional guidance</u> for information to include with your IRB application.



We will institute a data monitoring and safety plan. To mitigate and detect harm, the patient will be seen the week after surgery and again at six weeks. At these follow up visits, the PI will assess the subjects for any adverse events. The PI will assess for wound dehiscence, signs of infection, and necrosis. In addition, the patients will have access to the emergency contact information of Dr. Peter Timoney. The PI will be the sole monitor of the clinical investigation. Conflict of interest will be mitigated by comparing the surgeon's scar survey score to the patient's scar survey score. An independent group comprised of two or more non Study Personnel will review before/after photographs and scar surveys for acceptability. These photos and scar surveys will be stripped of identifiers prior to any non-study personnel reviewing. The group will prepare a summary report that will be submitted to the IRB.

If a significant discrepancy is apparent, we will not proceed onto the phase two. Toward this end, phase one of the protocol will investigate the scar phenotype of Dermabond closed wounds in a bilateral fashion so as to ascertain if there will be a significant difference between Dermabond and suture closed wounds. The results of phase 1 will be reported to the IRB after each datapoint is collected and the IRB will help decide if the study will proceed. We will not report events to any other entities besides the University of Kentucky ORI IRB. Any instance of wound dehiscence, necrosis or serious infection in the Dermabond group will be criteria for temporary suspension of the study. The development of any of these adverse effects in the superficial suture group will not result in study suspension.

Back to Top

# Future Use and Sharing of Material (e.g., Data/Specimens/Information)

If the material collected for this study will be used by members of the research team or shared with other researchers for future studies, please address the following:

- list the biological specimens and/or information that will be kept
- · briefly describe the types, categories and/or purposes of the future research
- · describe any risks of the additional use
- · describe privacy/confidentiality protections that will be put into place
- describe the period of time specimens/information may be used
- describe procedures for sharing specimens/information with secondary researchers
- · describe the process for, and limitations to, withdrawal of specimens/data



Are you recruiting or expect to enroll **Non-English Speaking Subjects or Subjects from a Foreign Culture**? (does not include short form use for incidentally encountered non-English subjects)

∩ Yes ∩ No

Non-English Speaking Subjects or Subjects from a Foreign Culture

#### **Recruitment and Consent:**

Describe how information about the study will be communicated to potential subjects appropriate for their culture, and if necessary, how new information about the research may be relayed to subjects during the study.

When recruiting Non-English-speaking subjects, provide a consent document in the subject's primary language. After saving this section, attach both the English and translated consent documents in the "Informed Consent" section.

# **Cultural and Language Consultants:**

The PI is required to identify someone who is willing to serve as the cultural consultant to the IRB.

- This person should be familiar with the culture of the subject population and/or be able to verify that translated documents are the equivalent of the English version of documents submitted.
- The consultant should not be involved with the study or have any interest in its IRB approval.
- Please include the name, address, telephone number, and email of the person who agrees to be the cultural consultant for your study.
- · ORI staff will facilitate the review process with your consultant. Please do not ask them to review your protocol separately.

For more details, see the IRB Application Instructions on Research Involving Non-English Speaking Subjects or Subjects from a Foreign Culture.

#### **Local Requirements:**

If you will conduct research at an international location, identify and describe:

- · relevant local regulations
- data privacy regulations
- · applicable laws
- ethics review requirements for human subject protection

Please provide links or sources where possible. If the project has been or will be reviewed by a local ethics review board, attach a copy in the "Additional Information/Materials" section. You may also consult the current edition of the <a href="International Compilation of Human Research Standards">International Compilation of Human Research Standards</a>

Does your study involve HIV/AIDS research and/or screening for other reportable diseases (e.g., Hepatitis c Yes © No

#### -HIV/AIDS Research

If you have questions about what constitutes a reportable disease and/or condition in the state of Kentucky, see ORI's summary sheet: "Reporting Requirements for Diseases and Conditions in Kentucky" [PDF].

**HIV/AIDS Research:** There are additional IRB requirements for designing and implementing the research and for obtaining informed consent. Describe additional safeguards to minimize risk to subjects in the space provided below.

For additional information, visit the online <u>IRB Survival Handbook</u> to download a copy of the "Medical IRB's requirements for Protection of Human Subjects in Research Involving HIV Testing" [D65.0000] [PDF], and visit the <u>Office for Human Research Protections web site</u> for statements on AIDS research, or contact the Office of Research Integrity at 859-257-9428.

## PI-Sponsored FDA-Regulated Research

Is this an investigator-initiated study that:

- 1) involves testing a Nonsignificant Risk (NSR) Device, or
- 2) is being conducted under an investigator-held Investigational New Drug (IND) or Investigational Device Exemption (IDE)? 
   Yes 
   No

#### PI-Sponsored FDA-Regulated Research

If the answer above is yes, then the investigator assumes the regulatory responsibilities of both the investigator and sponsor. The Office of Research Integrity provides a summary list of sponsor IND regulatory requirements for drug trials [PDF], IDE regulatory requirements for SR device trials [PDF], and abbreviated regulatory requirements for NSR device trials [PDF]. For detailed descriptions see FDA Responsibilities for Device Study Sponsors or FDA Responsibilities for IND Drug Study Sponsor-Investigators.

- Describe the experience/knowledge/training (if any) of the investigator serving as a sponsor (e.g., previously held an IND/IDE); and
- Indicate if any sponsor obligations have been transferred to a commercial sponsor, contract research organization (CRO), contract monitor, or other entity (provide details or attach FDA 1571).

Sponsor has completed multiple clinical trials in fellowship and as an attending.

IRB policy requires mandatory training for all investigators who are also FDA-regulated sponsors (see <a href="Sponsor-Investigator">Sponsor-Investigator</a> EAQs). A sponsor-investigator must complete the applicable Office of Research Integrity web based training, (drug or device) before final IRB approval is granted.

Has the sponsor-investigator completed the mandatory PI-sponsor training prior to this submission? ∘ Yes ○ No

If the sponsor-investigator has completed equivalent sponsor-investigator training, submit documentation of the content for the IRB's consideration.

# Attachments

| Attach Type | File Name |
|--------------------|----------------------|
| SponsorInvTraining | Timoney training.pdf |

HIPAA 0 unresolved comment(s)

Is HIPAA applicable? ⊙Yes ○No

(Visit ORI's <u>Health Insurance Portability and Accountability Act (HIPAA) web page</u> to determine if your research falls under the HIPAA Privacy Regulation.)

If yes, check below all that apply and attach the applicable document(s): 0

☐ HIPAA De-identification Certification Form

☐ HIPAA Waiver of Authorization

Attachments

# STUDY DRUG INFORMATION

0 unresolved comment(s)

# The term drug may include:

- FDA approved drugs,
- unapproved use of approved drugs,
- investigational drugs or biologics,
- other compounds or products intended to affect structure or function of the body, and/or
- complementary and alternative medicine products such as dietary supplements, substances generally recognized as safe (GRAS)
  when used to diagnose, cure mitigate, treat or prevent disease, or clinical studies of e-cigarettes examining a potential therapeutic
  purpose.

Does this protocol involve a drug including an FDA approved drug; unapproved use of an FDA approved drug; and/or an investigational drug?

If yes, complete the questions below. Additional study drug guidance.

| Non-Oncology). Use of IDS | is highly recommended, but option | Investigational Drug Service (IDS) pharmacies (Oncological for outpatient studies. Outpatient studies not using IDS pliance with drug accountability good clinical practices. |
|---|---|---|
| | ) will be housed and managed: | |
| | nvestigational Drug Service (IDS) UK Hospital | |
| Other Location: | | |
| la tha atudy baing canducto | d under a valid Investigational New | ( Drug (IND) application? |
| , , | d under a valid Investigational New | / Drug (IND) application? |
| C Yes C No | l complete the fallowing. | |
| If Yes, list IND #(s) and complete the following: | | |
| IND Submitted/Held by | <i>r</i> . | |
| IND Submitted/Held by | /:<br>Held By: | |
| Sponsor: □ | Held By: | |
| Sponsor: □ Investigator: □ | Held By: | |
| Sponsor: □ Investigator: □ Other: □ | Held By: Held By: | n's Expanded Access Program (e.g., Treatment IND) FDA Form 3926). |
| Sponsor: Investigator: Other: Checkmark if the stor if this is an Individu | Held By: Held By: Held By: udy is being conducted under FDA al Patient Expanded Access IND ( | |
| Sponsor: Investigator: Other: Checkmark if the stor if this is an Individual FDA's Expanded Accordillowing: FDA Form 3926 | Held By: Held By: Held By: udy is being conducted under FDA al Patient Expanded Access IND ( ess Program Information for Indivi | FDA Form 3926). dual Patient Expanded Access INDs, and attach the |
| Sponsor: Investigator: Other: Other: Checkmark if the stor if this is an Individual FDA's Expanded Accordillowing: FDA Form 3926 FDA expanded a | Held By: Held By: Held By: udy is being conducted under FDA al Patient Expanded Access IND (ess Program Information for Indivi | FDA Form 3926). dual Patient Expanded Access INDs, and attach the |

applicable drug documentation (e.g., Investigator Brochure; approved labeling; publication; FDA control of the document type.

Attachments

## STUDY DEVICE INFORMATION

0 unresolved comment(s)

## A DEVICE may be a:

- · component, part, accessory;
- · assay, reagent, or in-vitro diagnostic device;
- software, digital health, or mobile medical app;
- other instrument if intended to affect the structure or function of the body, diagnose, cure, mitigate, treat or prevent disease; or
- a homemade device developed by an investigator or other non-commercial entity and not approved for marketing by FDA.

For additional information, helpful resources, and definitions, see ORI's Use of Any Device Being Tested in Research web page.

Does this protocol involve testing (collecting safety or efficacy data) of a medical device including an FDA approved device, unapproved use of an approved device, humanitarian use device, and/or an investigational device?

Yes ○ No

[Note: If a marketed device(s) is only being used to elicit or measure a physiologic response or clinical outcome, AND, NO data will be collected on or about the device itself, you may answer "no" above, save and exit this section, (Examples: a chemo drug study uses an MRI to measure tumor growth but does NOT assess how effective the MRI is at making the measurement; an exercise study uses a heart monitor to measure athletic performance but no safety or efficacy information will be collected about the device itself, nor will the data collected be used for comparative purposes against any other similar device).]

If you answered yes above, please complete the following questions.

| Dermabond adhesive skin glue | |
|---|---|
| Is the study being conducted under a valid Investigational Device Exemption (IDE),<br>Humanitarian Device Exemption (HDE) or Compassionate Use? | |
| ດYes ເNo | |
| If Yes, complete the following: | |
| IDE or HDE #(s) | ·····g· |
| IDE/HDE Submitted/Hel | d by: |
| Sponsor: □ | Hold Du |
| · | Held By: |
| Investigator: □ | Held By: |
| Other: □ | Held By: |
| □ Check if this is a Tr | eatment IDE or Compassionate Use under the Food and Drug Administration (FDA) |
| Expanded Access pro | |
| | Group Expanded Access, see FDA's Early Expanded Access Program Information, |
| and attach the following: | |
| | cess approval or sponsor's authorization; |
| | sessment from an uninvolved physician, if available; reement from manufacturer or entity authorized to provide access to the product. |
| _ | |
| For guidance and reporting requirements at the conclusion of treatment see the Medical Device SOP. | |

Does the intended use of any research device being tested (not clinically observed) in this study meet the regul Significant Risk (SR) device?

- Yes. Device(s) being tested in this study presents a potential for serious risk to the health, safety, or welfare of a subject and (1) is intended as an implant; or (2) is used in supporting or sustaining human life; or (3) is of substantial importance in diagnosing, curing, mitigating or treating disease, or otherwise prevents impairment of human health; or (4) otherwise presents a potential for serious risk to the health, safety, or welfare of a subject.
- © No. All devices being tested in this study do not present a potential for serious risk to the health, safety, or welfare of subjects/participants.

Complete and attach the required <u>Study Device Form</u>, picking the "Study Device Form" for the document type. Any applicable device documentation (e.g., Manufacturer information; patient information packet; approved labeling; FDA correspondence, etc.) should be attached using "Other Device Documentation" for the document type.



# Attachments

| Attach Type | File Name |
|-------------------|------------------------------|
| Study Device Form | 77074_StudyDevice_335143.pdf |

# RESEARCH SITES

0 unresolved comment(s)

To complete this section, ensure the responses are accurate then click "SAVE".

A) Check all the applicable sites listed below at which the research will be conducted. If none apply, you do not need to check any boxes.

#### **UK Sites**

- □ UK Classroom(s)/Lab(s)

- □ UK Healthcare Good Samaritan Hospital
- □ UK Hospital

#### -Schools/Education Institutions

- □ Fayette Co. School Systems \*
- □ Other State/Regional School Systems
- □ Institutions of Higher Education (other than UK)

\*Fayette Co. School systems, as well as other non-UK sites, have additional requirements that must be addressed. See ORI's <u>IRB Application Instructions - Off-site Research</u> web page for details.

## Other Medical Facilities

- □ Bluegrass Regional Mental Health Retardation Board
- □ Cardinal Hill Hospital
- □ Eastern State Hospital
- □ Norton Healthcare
- □ Nursing Homes
- ☐ Shriner's Children's Hospital
- □ Veterans Affairs Medical Center
- □ Other Hospitals and Med. Centers
- □ Correctional Facilities
- □ Home Health Agencies
- □ International Sites

Research activities conducted at performance sites that are not owned or operated by the University of Kentucky (UK) or at sites that do not fall under the UK IRB's authority, are subject to special procedures for coordination of research review. Additional information is required (see IRB Application Instructions - Off-Site Research web page), including:

- A letter of support and local context is required from non-UK sites. See *Letters of Support and Local Context* on the IRB Application Instructions Off-Site Research web page for more information.
- Supportive documentation, including letters of support, can be attached below.
- NOTE: If the non-UK sites or non-UK personnel are engaged in the research, there are additional federal and
  university requirements which need to be completed for their participation. For instance, the other site(s) may need
  to complete their own IRB review, or a cooperative review arrangement may need to be established with non-UK
  sites.

 Questions about the participation of non-UK sites/personnel should be discussed with the ORI staff 9428.

List all other non-UK owned/operated locations where the research will be conducted:

Describe the role of any non-UK site(s) or non-UK personnel who will be participating in your research.

Attachments

B) Is this a multi-site study for which you are the lead investigator or UK is the lead site? Yes No

If YES, describe the plan for the management of reporting unanticipated problems, noncompliance, and submission of protocol modifications and interim results from the non-UK sites:

C) If your research involves collaboration with any sites and/or personnel outside the University of Kentucky, then it is considered multisite research and IRB reliance issues will need to be addressed. This may include national multi-center trials as well local studies involving sites/personnel external to UK. If you would like to request that the University of Kentucky IRB (UK IRB) serve as the lead IRB for your study, or if you would like the UK IRB to defer review to another IRB, please contact the <a href="mailto:IRBReliance@uky.edu">IRBReliance@uky.edu</a>.
#### **RESEARCH ATTRIBUTES**

0 unresolved comment(s)

Indicate the items below that apply to your research. Depending on the items applicable to your research, you may be required to complete additional forms or meet additional requirements. Contact the ORI (859-257-9428) if you have questions about additional requirements.

□ Not applicable

## -Check All That Apply-

- □ Academic Degree/Required Research
- □ Alcohol/Drug/Substance Abuse Research
- □ Biological Specimen Bank Creation (for sharing)
- □ Cancer Research
- CCTS-Center for Clinical & Translational Science
- □ Certificate of Confidentiality
- □ Clinical Research
- □ Clinical Trial Phase 1
- □ Collection of Biological Specimens for internal banking and use (not sharing)
- ☐ Community-Based Participatory Research
- □ Deception
- □ Educational/Student Records (e.g., GPA, test scores)
- □ Emergency Use (Single Patient)
- □ Gene Transfer
- ☐ Genetic Research
- $\hfill \square$  GWAS (Genome-Wide Association Study) or NIH Genomic Data Sharing (GDS)
- □ Human Cells, Tissues, and Cellular and Tissue Based Products
- □ Individual Expanded Access or Compassionate Use
- □ International Research
- □ Planned Emergency Research Involving Exception from Informed Consent
- □ Recombinant DNA
- □ Registry or data repository creation
- ☐ Stem Cell Research
- ☐ Suicide Ideation or Behavior Research
- □ Survey Research
- □ Transplants
- $\hfill\Box$  Use, storage and disposal of radioactive material and radiation producing devices
- □ Vaccine Trials

For additional requirements and information:

- Cancer Research (MCC PRMC)
- Certificate of Confidentiality (look up "Confidentiality/Privacy...")
- CCTS (Center for Clinical and Translational Science)
- <u>Clinical Research</u> (look up "What is the definition of....)
- Clinical Trial
- Collection of Biological Specimens for Banking (look up "Specimen/Tissue Collection...")
- <u>Collection of Biological Specimens</u> (look up "Specimen/Tissue Collection...")
- Community-Based Participatory Research (look up "Community-Engaged...")
- Data & Safety Monitoring Board (DSMB)

\*For Medical IRB: <u>Service Request Form</u> for CCTS DSMB

- Data & Safety Monitoring Plan
- Deception\*

\*For deception research, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"

- Emergency Use (Single Patient) [attach Emergency Use Checklist] (PDF)
- Genetic Research (look up "Specimen/Tissue Collection...")
- Gene Transfer
- <u>HIV/AIDS Research</u> (look up "Reportable Diseases/Conditions")
- Screening for Reportable Diseases [E2.0000] (PDF)
- International Research (look up "International & Non-English Speaking")
- NIH Genomic Data Sharing (GDS) Policy (PDF)
- Planned Emergency Research Involving Waiver of Informed Consent\*

\*For Planned Emergency Research Involving Waiver of Informed Consent, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"

• <u>Use, storage and disposal of radioactive material</u> <u>and radiation producing devices</u>

# FUNDING/SUPPORT

0 unresolved comment(s)

If the research is being submitted to, supported by, or conducted in cooperation with an external or internal agency or funding program, indicate below all the categories that apply. ①

Not applicable

#### -Check All That Apply

- □ Grant application pending
- (HHS) Dept. of Health & Human Services
- (NIH) National Institutes of Health
- $\ \ \square$  (CDC) Centers for Disease Control & Prevention
- □ (HRSA) Health Resources and Services
   Administration

- Federal Agencies Other Than Those Listed Here
- Industry (Other than Pharmaceutical Companies)
- Internal Grant Program w/ proposal
- Internal Grant Program w/o proposal
- National Science Foundation
- Other Institutions of Higher Education
- Pharmaceutical Company
- □ Private Foundation/Association
- **■** U.S. Department of Education

Other:

Click applicable listing(s) for additional requirements and information:

- (HHS) Dept. of Health & Human Services
- (NIH) National Institutes of Health
- (CDC) Centers for Disease Control & Prevention
- (HRSA) Health Resources & Services Administration
- (SAMHSA) Substance Abuse & Mental Health Services Administration
- Industry (Other than Pharmaceutical Companies) [IRB Fee Info]
- National Science Foundation
- (DoEd) U.S. Department of Education
- (DoJ) Department of Justice or Bureau of Prisons
- (DoE) Department of Energy Summary and Department of Energy Identifiable Information Compliance Checklist
- (EPA) Environmental Protection Agency

Specify the funding source and/or cooperating organization(s) (e.g., National Cancer Institute, Ford Foundation, Eli Lilly & Company, South Western Oncology Group, Bureau of Prisons, etc.):

#### Add Related Grants

If applicable, please search for and select the OSPA Account number or Electronic Internal Approval Form (eIAF) # (notif #) associated with this IRB application using the "Add Related Grants" button.

If required by your funding agency, upload your grant using the "Grant/Contract Attachments" button.

Add Related Grants

**Grant/Contract Attachments** 

The research involves use of Department of Defense (DoD) funding, military personnel, DoD facilities, or other DoD resources. (See <u>DoD SOP</u> and <u>DoD Summary</u> for details)

Yes 
 No

Using the "attachments" button (below), attach applicable materials addressing the specific processes described in the DoD SOP.

DOD SOP Attachments

Additional Certification: (If your project is federally funded, your funding agency may request an Assurance/ Certification/Deform.) Check the following if needed:

□ Protection of Human Subjects Assurance/Certification/Declaration of Exemption (Formerly Optional Form – 310)

Assurance/Certification Attachments

#### **OTHER REVIEW COMMITTEES**

0 unresolved comment(s)

If you check any of the below committees, additional materials may be required with your application submission.

Does your research fall under the purview of any of the other review committees listed below? [If yes, check all that apply and attach applicable materials using the attachment button at the bottom of your screen.]

∩ Yes ⊙ No

#### **Additional Information**

- □ Institutional Biosafety Committee
- □ Radiation Safety Committee
- ☐ Radioactive Drug Research Committee
- ☐ Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC)
- ☐ Graduate Medical Education Committee (GME)
- ☐ Office of Medical Education (OME)
- Institutional Biosafety Committee (IBC) Attach required IBC materials
- Radiation Safety Committee (RSC) For applicability, see instructions and attach form
- Radioactive Drug Research Committee (RDRC)
- Markey Cancer Center (MCC) Protocol Review and Monitoring <u>Committee (PRMC)\*\*\*</u> - Attach MCC PRMC materials, if any, per instructions.
- Office of Medical Education (OME)
- Graduate Medical Education Committee (GME)

# Attachments

\*\* If your study involves cancer research, be sure to select "Cancer Research" in the "Research Attributes" section. ORI will send your research protocol to the Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC). The MCC PRMC is responsible for determining whether the study meets the National Cancer Institute (NCI) definition of a clinical trial and for issuing documentation to you (the investigator) which confirms either that PRMC approval has been obtained or that PRMC review is not required. Your IRB application will be processed and reviewed independently from the PRMC review.

#### ADDITIONAL INFORMATION/MATERIALS

0 unresolved comment(s)

Do you want specific information inserted into your approval letter? c Yes 6 No

Approval Letter Details:

If you wish to have specific language included in your approval letter (e.g., serial #, internal tracking identifier, etc...), type that language in the box below exactly as it should appear in the letter. The text you enter will automatically appear at the top of all approval letters, identical to how you typed it, until you update it. Don't include instructions or questions to ORI staff as those will appear in your approval letter. If these details need to be changed for any reason, you are responsible for updating the content of this field.

#### Additional Materials:

If you have other materials you would like to include for the IRB's consideration, check all that apply and attach the corresponding documents using the Attachments button below.

- □ Detailed protocol
- □ Dept. of Health & Human Services (DHHS) approved protocol (such as NIH sponsored Cooperative Group Clinical Trial)
- □ Other Documents

Protocol/Other Attachments

Attach Type File Name
Other IRB Requested Revisions.pdf

NOTE: Instructions for Dept. of Health & Human Services (DHHS)-approved protocol

If you have password protected documents, that feature should be disabled prior to uploading to ensure access for IRB review.

To view the materials currently attached to your application, click "All Attachments" on the left menu bar.

## **SIGNATURES (ASSURANCES)**

0 unresolved comment(s)

#### Introduction

All IRB applications require additional assurances by a Department Chairperson or equivalent (DA), and when applicable, a Faculty Advisor or equivalent (FA). This signifies the acceptance of certain responsibilities and that the science is meritorious and deserving of conduct in humans. The person assigned as DA should not also be listed in the Study Personnel section, and the individual assigned as FA should be listed in the Study Personnel section.

For a list of responsibilities reflected by signing the Assurance Statement, refer to "What does the Department Chairperson's Assurance Statement on the IRB application mean?"

For a detailed illustration of how to complete this section, please review the short online video tutorial "Signatures (Assurance) Section - How to Complete." Otherwise, follow the steps below.

# **Required Signatures:**

| 0 | | | | | |
|---|---|---|---|---|---|
| First<br>Name | Last<br>Name | Role | Department | Date<br>Signed | |
| Paul | Pearson | Department<br>Authorization | Ophthalmology<br>& Visual<br>Science | 06/08/2023<br>06:48 AM | View/Sign |
| Peter | Timoney | Principal<br>Investigator | Ophthalmology<br>& Visual<br>Science | 06/08/2023<br>11:53 AM | View/Sign |

#### Department Authorization

r This is to certify that I have reviewed this research protocol and that I attest to the scientific validity and importance of this study; to the qualifications of the investigator(s) to conduct the project and their time available for the project; that facilities, equipment, and personnel are adequate to conduct the research; and that continued guidance will be provided as appropriate. When the principal investigator assumes a sponsor function, the investigator has been notified of the additional regulatory requirements of the sponsor and by signing the principal investigator Assurance Statement, confirms he/she can comply with them.

\*If the Principal Investigator is also the Chairperson of the department, the Vice Chairperson or equivalent should complete the "Department Authorization".

\*\*IF APPLICABLE FOR RELIANCE: I attest that the principal investigator has been notified of the regulatory requirements of both the Reviewing and Relying IRBs, according to the information provided in the E-IRB application. The attached Reliance Assurance Statement, signed by the principal investigator, confirms that he/she can comply with both sets of IRB requirements.

#### Principal Investigator's Assurance Statement

I understand the University of Kentucky's policies concerning research involving human subjects and I agree:

- 1. To comply with all IRB policies, decisions, conditions, and requirements;
- 2. To accept responsibility for the scientific and ethical conduct of this research study;
- 3. To obtain prior approval from the Institutional Review Board before amending or altering the research protocol or implementing changes in the approved consent/assent form;
- 4. To report to the IRB in accord with IRB/IBC policy, any adverse event(s) and/or unanticipated problem(s) involving risks to subjects;
- 5. To complete, on request by the IRB for Full and Expedited studies, the Continuation/Final Review Forms;
- 6. To notify the Office of Sponsored Projects Administration (OSPA) and/or the IRB (when applicable) of the development of any financial interest not already disclosed;
- 7. Each individual listed as study personnel in this application has received the mandatory human research protections

- education (e.g., CITI);
- 8. Each individual listed as study personnel in this application possesses the necessary experience for conducting research activities in the role described for this research study.
- 9. To recognize and accept additional regulatory responsibilities if serving as both a sponsor and investigator for FDA regulated research.

Furthermore, by checking this box, I also attest that:

- I have appropriate facilities and resources for conducting the study;
- I am aware of and take full responsibility for the accuracy of all materials submitted to the IRB for review;
- If applying for an exemption, I also certify that the only involvement of human subjects in this research study will be in the categories specified in the Protocol Type: Exemption Categories section.
- If applying for an Abbreviated Application (AA) to rely on an external IRB, I understand that certain items above (1, 3, 4, 7-8) may not apply, or may be altered due to external institutional/IRB policies. I document my agreement with the <a href="Principal Investigator Reliance Assurance Statement">Principal Investigator Reliance Assurance Statement</a> by digitally signing this application.

\*You will be able to "sign" your assurance after you have sent your application for signatures (use Submission section). Please notify the personnel required for signing your IRB application after sending for signatures. Once all signatures have been recorded, you will need to return to this section to submit your application to ORI.

#### SUBMISSION INFORMATION

0 unresolved comment(s)

\*\*\* If this Continuation Review entails a change in the scope of your activities to include COVID-19 related research, please insert "COVID19" at the start of your Project and Short Titles.\*\*\*

Each Section/Subsection in the menu on the left must have a checkmark beside it (except this Submission section) indicating the Section/Subsection has been completed. Otherwise your submission for IRB review and approval cannot be sent to the Office of Research Integrity/IRB.

If applicable, remember to update the Approval Letter Details text box under the Additional Information section

If your materials require review at a convened IRB meeting which you will be asked to attend, it will be scheduled on the next available agenda and you will receive a message to notify you of the date.

If you are making a change to an attachment, you need to delete the attachment, upload a highlighted version that contains the changes (use Document Type of "Highlighted Changes"), and a version that contains the changes without any highlights (use the appropriate Document Type for the item(s)). Do **not** delete approved attachments that are still in use.

-Principal Investigator's Assurance Statement

I understand the University of Kentucky's policies concerning research involving human subjects, and I attest to:

- 1. Having reviewed all the investigational data from this study, including a compilation of all internal and external unanticipated problems.
- 2. Having reviewed, if applicable, information from the sponsor including updated investigator brochures and data and safety monitoring board reports.

I also attest that I have reviewed pertinent materials concerning the research and concluded:

• The human subject risk/benefit relationship is unaffected, mitigated, or eliminated by closure of the study and all pertinent materials for closure of the research are being submitted to the IRB for consideration.

■ By checking this box, I am providing assurances for the applicable items listed above.

Your protocol has been submitted.

# Download all

| | Document Type | File Loaded | Document<br>Description | File<br>Size | Modified<br>By | Mod Date |
|---|---|---|---|---|---|---|
| 4 | StudyClosure | StudyClosure.pdf | | 0.079 | jlkear0 | 6/20/2024 8:34:11<br>AM |
| 4 | CR_EntireConsent | Patient 7 Consent.pdf | | 5.986 | ccbl229 | 6/2/2024 11:30:22<br>PM |
| 4 | CR_EntireConsent | Patient 6 consent.pdf | | 3.148 | ccbl229 | 6/2/2024 11:30:12<br>PM |
| 4 | StudyDevice | 77074_StudyDevice_335143.pdf | | 1.050 | ccbl229 | 7/26/2023 2:58:04<br>PM |
| 4 | SponsorInvTraining | Timoney training.pdf | | 0.062 | ccbl229 | 7/25/2023 3:11:50<br>PM |
| 4 | AddInfoProduct | IRB Requested Revisions.pdf | IRB Requested Revisions | 0.242 | scbe223 | 7/11/2023 3:49:02<br>PM |
| 4 | DataCollection | dss_2017_12_22_patel_ds-00686-<br>2016_sdc1.pdf | POSAS observer scale | 0.119 | ccbl229 | 6/7/2023 11:28:05<br>PM |
| 4 | DataCollection | 77074_DataCollection_267377.pdf | Scar Survey | 0.169 | ccbl229 | 6/7/2023 11:12:45<br>PM |

**Protocol Changes** 

Protocol Nu.

88617 CLOSED

Click link to sort Changed Date
Project Information IsRelianceRequested changed by ccbl229 on 6/2/2024 11:24:52 PM
N

Study Personnel Changes:

#### Protocol Type Comment by Cody Blanchard - PI to PI on 6/4/2024 3:45:54 PM

Hi, this question does not apply to our study. There were no results to communicate as there were no tests that were done. This was purely an observational study with a survey that the patient filled out in their postop appointment. I am not sure what the violation is that is being alleged here

Protocol Type Comment by Jennifer Kearns - ORI to IRB/PI on 6/4/2024 3:03:53 PM

Both of the uploaded signed consents are missing checkboxes and initials in the paragraph re: permission to contact participants for return of results or incidental findings (p. 4.). Please submit a violation report for this issue and include the following: 1) Was this missed on all of the signed consents? and 2) Do you anticipate any issues arising from missing this selection? (i.e., how likely is it that there were any incidental findings or results to be returned?) Let me know if you have questions about this request.

Date: March 30, 2025

Identifiers: NCT05981443 Unique Protocol ID: BrowPtosis

Brief An Analysis of Dermabond vs. Non-Absorbable Sutures in Skin Closure for

Title: Brow Ptosis Procedures

Our statistical analysis plan for this pilot study consists of using only data gathered using the POSAS survey administered to patients at their post-operative visits. We used this survey and demographic data to perform basic descriptive statistics to detect if there was a difference between the reported rates of patient satisfaction and ratings of their scars.



# Consent and Authorization to Participate in a Research Study

# KEY INFORMATION FOR SCAR ANALYSIS IN DIRECT EXCISION BROW LIFT: COMPARING OCTYL-2-CYANOACRYLARTE (DERMABOND) VERSUS NON-ABSORBABLE SUTURES

We are asking you to choose whether or not to volunteer for a research study about scar appearance after brow lift surgery. We are asking you because you may receive this brow lift surgery soon. This page is to give you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

# WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

By doing this study, we hope to learn about scar formation differences between two commonly used surgical closing techniques. The device being evaluated is Dermabond, which is used for skin closure in many different medical procedures but is investigational in brow ptosis, versus the standard of care, which is non-absorbable sutures. Your participation in this research will last about 3 months. You will fill out a survey about the appearance of your scar 10 days and 3 months after surgery.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

To help us understand the nature of scar formation between these two common surgical methods for closing skin. For a complete description of benefits, refer to the Detailed Consent.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

Reasons to not participate in this study is that it will not directly benefit your health and you will be randomly assigned to a procedure group. For a complete description of risks, refer to the Detailed Consent.

An alternative to participating in this study is to not participate. For a complete description of alternate treatment/procedures, refer to the Detailed Consent.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

As a student, if you decide not to take part in this study, your choice will have no effect on your academic status or class grade(s).

# WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study contact Peter Timoney, MD, of the University of Kentucky, Department of Ophthalmology at 859 218 2609.

If you have any concerns or questions about your rights as a volunteer in this research, contact staff in the University of Kentucky (UK) Office of Research Integrity (ORI) between the business hours of 8am and 5pm EST, Monday-Friday at 859-257-9428 or toll free at 1-866-400-9428.

## **DETAILED CONSENT:**

#### ARE THERE REASONS WHY YOU WOULD NOT QUALIFY FOR THIS STUDY?

If you are under the age of 18 or older the age of 100, you will not quality for this study. In addition, if you are only receiving a brow lift on one side, you will not qualify.

#### WHERE WILL THE STUDY TAKE PLACE AND WHAT IS THE TOTAL AMOUNT OF TIME INVOLVED?

The research procedures will be conducted at the University of Kentucky Department of Ophthalmology Clinics. You will need to come to two short follow up visits during the study (one week after the surgery and 2-3 months afterwards) and complete one survey from home.

## WHAT WILL YOU BE ASKED TO DO?

Eligible subjects will be asked to undergo one of two different skin closing techniques for their brow ptosis (heavy or droopy eyes) repair. Subjects will be randomly assigned to a treatment arm of right brow vs. left brow using a computer generator. The skin closing techniques are all in common use and considered normal care. The first technique is using sutures to close the outer most part of your eyelid skin. The second technique uses Dermabond (skin adhesive glue) to close the outer most part of your eyelid skin. All other aspects of the procedure are the same. Dermabond is not routinely used at University of Kentucky during brow lift procedures for closure of outer most part of the eyelid skin, but Dermabond is FDA approved for closure of wounds from minimally invasive surgery. Subsequently, you will complete a survey to grade the appearance of each scar. Before and after photographs will also be taken for research purposes.

# WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

One possible risk is the formation of scars. While the surgical glue is commonly used to close small wounds (like those in your procedure), there is limited experience in using it in this particular surgery. Any wound closure is subject to infection and wound dehiscence (wound opening). Another risk that is possible but unlikely is a local skin reaction to the Dermabond.

In the case of a breach in confidentiality, your social, psychological, and emotional health may be put at risk.

There is always a chance that any medical treatment can harm you. The research treatments/procedures in this study are no different. In addition to risks described in this consent, you may experience a previously unknown risk or side effect.

# WILL YOU BENEFIT FROM TAKING PART IN THIS STUDY?

You will not get any personal benefit from taking part in this study.

## IF YOU DON'T WANT TO TAKE PART IN THE STUDY, ARE THERE OTHER CHOICES?

If you do not want to be in the study, there are no other choices except not to take part in the study. Your standard of care will not be affected by choosing not to participate.

## WHAT WILL IT COST YOU TO PARTICIPATE?

There is no additional cost for participation in this study.

You and/or your insurance company, Medicare, or Medicaid will be responsible for the costs of all care and treatment that you would normally receive for any conditions you may have. These are costs that are considered medically necessary and will be part of the care you receive even if you do not take part in this study.

The University of Kentucky may not be allowed to bill your insurance company, Medicare, or Medicaid for the medical

procedures done strictly for research. Therefore, these costs will be paid by the study.

#### WHO WILL SEE THE INFORMATION THAT YOU GIVE?

When we write about or share the results from the study, we will write about the combined information. We will keep your name and other identifying information private. We will make every effort to prevent anyone who is not on the research team from knowing that you gave us information, or what that information is. We will make every effort to prevent anyone who is not on the research team from accessing your information or knowing your status in the study. In order to protect the confidentiality of our data, we will utilize the following tactics: remove identifying information (i.e. name) from medical information; store medical information in a password-protected database; and limit access to view medical information to the research team who sign a law-binding contract to not divulge any information. When transporting any medical information on a portable storage device, any and all portable storage devices will be encrypted and require a password to access. Any paper records used to record data will be shredded or disposed in a patient information protected manner after the data is recorded on an electronic system.

You should know that in some cases we may have to show your information to other people because

For example, the law may require us to share your information with:

- a court or agencies, if you have a reportable disease/condition;
- authorities, if you report information about a child being abused; or if you pose a danger to yourself or someone else.

REDCap is a secure, web-based program to capture and store data at the University of Kentucky. We will make every effort to safeguard your data in REDCap. However, given the nature of online surveys, we cannot guarantee the security of data obtained by way of the Internet.

#### CAN YOU CHOOSE TO WITHDRAW FROM THE STUDY EARLY?

You can choose to leave the study at any time. You will not be treated differently if you decide to stop taking part in the study.

If you choose to leave the study early, data collected until that point will remain in the study database and may not be removed.

The investigators conducting the study may need to remove you from the study. You may be removed from the study if:

- you are not able to follow the directions,
- we find that your participation in the study is more risk than benefit to you, or

# ARE YOU PARTICIPATING, OR CAN YOU PARTICIPATE, IN ANOTHER RESEARCH STUDY AT THE SAME TIME AS PARTICIPATING IN THIS ONE?

You may take part in this study if you are currently involved in another research study. It is important to let the investigator/your doctor know if you are in another research study. You should discuss this with the investigator/your doctor before you agree to participate in another research study while you are in this study.

# WHAT HAPPENS IF YOU GET HURT OR SICK DURING THE STUDY?

If you believe you are hurt or if you get sick because of something that is due to the study, you should call Peter Timoney, M.D. at (859 218 2609) immediately.

Dr. Peter Timoney will determine what type of treatment, if any, is best for you at that time.

It is important for you to understand that the University of Kentucky does not have funds set aside to pay for the cost of any care or treatment that might be necessary because you get hurt or sick while taking part in this study. Also, the University of Kentucky will not pay for any wages you may lose if you are harmed by this study.

Medical costs related to your care and treatment because of study-related harm.

will be your responsibility

You do not give up your legal rights by signing this form.

# WILL YOU RECEIVE ANY REWARDS FOR TAKING PART IN THIS STUDY?

You will not receive any rewards or payment for taking part in the study.

# WHAT IF NEW INFORMATION IS LEARNED DURING THE STUDY THAT MIGHT AFFECT YOUR DECISION TO PARTICIPATE?

We will tell you if we learn new information that could change your mind about staying in the study. We may ask you to sign a new consent form if the information is provided to you after you have joined the study.

## WILL YOU BE GIVEN INDIVIDUAL RESULTS FROM THE RESEARCH TESTS?

| Generally, tests done for research purposes are not meant to provide clinical information. We will not provide you with individual research results. | | | |
|---|---|---|---|
| be important to y | you/your family | | sults or incidental findings that are determined to<br>e unforeseen findings discovered during the<br>lth). |
| □ Ye | es 🗆 No | Initials | |
| You may also withdraw your consent to be contacted with information about research results or incidental findings by sending a written request to ATTN: Peter Timoney, MD 110 Conn Terrace, Suite 550 Lexington, KY 40508. | | | |
| WILL WE CONTACT YOU WITH INFORMATION ABOUT PARTICIPATING IN FUTURE STUDIES? | | | |
| The research staff would like to contact you in the future with information about participating in additional studies. If so, it will be limited to 2 times per year. | | | |
| Do you give your permission to be contacted in the future by Dr. Timoney or his staff regarding your willingness to participate in future research studies? | | | |

# WHAT ELSE DO YOU NEED TO KNOW?

If you volunteer to take part in this study, you will be one of 10 people to do so at the University of Kentucky.

# WILL YOUR INFORMATION BE USED FOR FUTURE RESEARCH?

Your information collected for this study will NOT be used or shared for future research studies, even if we remove the identifiable information like your name, medical record number, or date of birth.

#### AUTHORIZATION TO USE OR DISCLOSE YOUR IDENTIFIABLE HEALTH INFORMATION

The privacy law, HIPAA (Health Insurance Portability and Accountability Act), requires researchers to protect your health information. The following sections of the form describe how researchers may use your health information.

# Your health information that may be accessed, used and/or released includes:

Demographic information and scar survey results. Demographic information includes age, sex, and race.
 Patient history and physical exam findings may be reported in a scientific journal article.

# The Researchers may use and share your health information with:

- The University of Kentucky's Institutional Review Board/Office of Research Integrity;
- Law enforcement agencies when required by law;
- University of Kentucky representatives;
- RedCaps online secure survey platform
- FDA (Food and Drug Administration)
- UK Health System (EPIC, the electronic medical record)
- Health Systems outside of UK with which you have a patient relationship

The researchers agree to only share your health information with the people listed in this document.

Should your health information be released to anyone that is not regulated by the privacy law, your health information may be shared with others without your permission; however, the use of your health information would still be regulated by applicable federal and state laws.

You may not be allowed to participate in the research study if you do not sign this form. If you decide not to sign this form, it will not affect your:  $\tilde{\varphi}'$ 

- Current or future healthcare at the University of Kentucky;
- Current or future payments to the University of Kentucky;
- · Ability to enroll in any health plans (if applicable); or
- Eligibility for benefits (if applicable).

After signing the form, you can change your mind and NOT let the researcher(s) collect or release your health information (revoke the Authorization). If you revoke the authorization:

- Send a written letter to: Peter Timoney at 110 Conn Terrace, Suite 550 Lexington, KY 40508 to inform him of your decision.
- Researchers may use and release your health information **already** collected for this research study.
- Your protected health information may still be used and released should you have a bad reaction (adverse event).

The use and sharing of your information has no time limit.

If you have not already received a copy of the Privacy Notice, you may request one. If you have any questions about your privacy rights, you should contact the University of Kentucky's Privacy Officer between the business hours of 8am and 5pm EST, Monday-Friday at (859) 323-1184.

# **Appendix: Scar Survey**

# **POSAS Patient scale**

| The Patient and Observer Scar Assessment Scale v2.0 / EN Date of examination: Name of pa | tient: | |
|---|---|---|
| Observer: | | |
| Location: Date of birth | h: | |
| Research / study: Identification | on number: | |
| | 1 = no, not at all 1 2 3 4 5 | yes, very much = 10 6 7 8 9 10 |
| HAS THE SCAR BEEN PAINFUL THE PAST FEW WEEKS? | 00000 | |
| HAS THE SCAR BEEN ITCHING THE PAST FEW WEEKS? | | |
| TABLE. | 0000 | |
| | 1 = no, as normal skin | yes, very different = 10 |
| | 1 = no, as normal skin | yes, very different = 10 |
| S THE SCAR COLOR DIFFERENT FROM THE COLOR OF YOUR NORMAL SKIN AT PRESENT? | 1 = no, as normal skin | yes, very different = 10 |
| S THE SCAR COLOR DIFFERENT FROM THE COLOR OF YOUR NORMAL SKIN AT PRESENT? S THE STIFFNESS OF THE SCAR DIFFERENT FROM YOUR NORMAL SKIN AT PRESENT? | 1 = no, as normal skin | yes, very different = 10 |
| IS THE SCAR COLOR DIFFERENT FROM THE COLOR OF YOUR NORMAL SKIN AT PRESENT? IS THE STIFFNESS OF THE SCAR DIFFERENT FROM YOUR NORMAL SKIN AT PRESENT? IS THE THICKNESS OF THE SCAR DIFFERENT FROM YOUR NORMAL SKIN AT PRESENT? IS THE SCAR MORE IRREGULAR THAN YOUR NORMAL SKIN AT PRESENT? | 1 = no, as normal skin | yes, very different = 10 |

# INFORMED CONSENT SIGNATURES

| This consent includes the following |
|-------------------------------------|
|-------------------------------------|

- Key Information Page
- Detailed Consent
- Scar Survey

You will receive a copy of this consent form after it has been signed.

| Signature of research subject | Date | |
|---|---|---|
| Printed name of research subject | | |
| Printed name of [authorized] person obtaining informed consent and HIPAA authorization | | <br>Date |